CLINICAL TRIAL: NCT00599625
Title: Pravastatin Therapy in Patients With Active Crohn's Disease: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Brian Behm, MD, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11453
Record Dates: First submitted 2007-12-26; First posted 2008-01-24 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients with active Crohn's Disease
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — 80mg administered daily for 6 consecutive weeks

SUMMARY:
The primary objective of this study is to provide data regarding clinical and immunologic activity of oral doses of pravastatin 80mg administered daily for 6 consecutive weeks, for the treatment of active Crohn's disease as shown by the Harvey-Bradshaw Index (HBI) and/or elevated C-reactive protein (CRP).

We hypothesize pravastatin will significantly reduce symptoms of Crohn's disease, as shown by a decrease in HBI, by the end of the study period. Secondary outcomes of this study include the effect of pravastatin on C-reactive protein, ESR, proinflammatory cytokines, and fecal lactoferrin.

DETAILED DESCRIPTION:
The HMG CoA (3-hydroxy-3-methylglutarylcoenzyme A) reductase inhibitors (statins) have been found to significantly reduce cardiovascular morbidity and mortality (1,2). While these clinical benefits are mediated in part by changes in lipids, particularly reductions in low-density lipoproteins (LDL), recent studies have suggested broader anti-inflammatory effects may also play a role by modifying various inflammatory pathways (3). Statins inhibit the synthesis of several proinflammatory cytokines, including tumor necrosis factor-alpha (TNF-alpha), IL-6, and IL-8 (4,5). Statins have also been shown to reduce inflammation by down regulating expression of MHC II molecules (6). Statins inhibit the production of chemokines and C-reactive protein (CRP), both molecules involved in inflammation (7-9).

On the basis of this data, several investigators have evaluated the effects of statin therapy in several inflammatory diseases. Recent studies evaluating inflammatory arthritis found that statins significantly decreased inflammation in an animal model (10). Statins also appear to reduce the severity of chemically induced peritonitis in rats, primarily by interfering with leukocyte adhesion and extravasation (11).

In humans, two small studies evaluating the use of statins in patients with rheumatoid arthritis and several other autoimmune diseases found that short-term use of statins was associated with significant decreases in disease activity and biochemical markers of inflammation (12,13). A subsequent randomized, double-blinded study evaluating the role of atorvastatin in 116 patients with rheumatoid arthritis found significant reductions in the number of swollen joints and levels of several markers of inflammation, including ESR and CRP, after 6 months of therapy compared with placebo (14). This animal and human data confirm HMG CoA-reductase inhibitors play a role in modulating inflammatory pathways, and suggest statins may have significant therapeutic potential in a range of chronic inflammatory diseases.

The use of pravastatin has been shown to inhibit the development of colitis in a rat model (15). Dextran sulfate (DSS) is a chemical that causes intestinal injury when given enterally to animals, and DSS-induced colitis has been found to share many characteristics with inflammatory bowel disease. Rats given DSS typically become cachectic, develop hematochezia, and develop abnormalities of intestinal epithelial permeability. Rats do not develop intestinal injury when DSS is given concomitantly with pravastatin. Pravastatin appears to prevent intestinal injury at least in part by increased eNOS expression, which is typically degraded by DSS administration (15). This animal model suggests that statins could potentially play a role in reducing the inflammation associated with active inflammatory bowel disease, and could potentially be a safe and well tolerated adjunctive therapy for the treatment of inflammatory bowel disease.

This study is an open label pilot study designed to assess the safety and efficacy of pravastatin on patients with active Crohn's disease. Patients enrolled in the study will be given pravastatin 80mg daily for a total of six weeks. The primary endpoint will be reduction in clinical disease activity, as measured by the Harvey-Bradshaw Index (HBI). Patients will also be assessed for biochemical markers of inflammation before and at completion of the study to assess the impact of pravastatin on these markers.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females on an adequate contraceptive regimen aged 18-65
* Active Crohn's disease (HBI >5 or serum CRP concentration above the upper limits of normal on initial labs.
* Stable regimen of medications for treatment of Crohn's disease for at least 4 weeks and will continue the current regimen for the 6 weeks of drug administration. Patients taking azathioprine/6-MP and methotrexate will need to be on a stable dose of these medications for a minimum of 8 weeks prior to study enrollment.
* Medications for the treatment of Crohn's disease meeting inclusion criteria are azathioprine/6-MP, methotrexate, mesalamine, ciprofloxacin, metronidazole, budesonide, and/or less than or equal to 20mg prednisone or an equivalent steroid per day

Exclusion Criteria:

* Patients less than 18 or greater than 65
* Current therapy with a statin or alternative medication for hyperlipidemia
* Hypersensitivity or known adverse reaction to statin therapy in the past
* Pregnancy
* Use of cyclosporin, erythromycin, and/or greater than 20mg of prednisone or its equivalent per day during the 4 weeks prior to study entry and/or during the 6 week study drug administration period.
* Use of infliximab during 8 weeks prior to study entry and/or during the 6 week study drug administration period.
* AST, ALT or CK more than twice the upper limits of normal on baseline laboratory data
* Serum creatinine greater than 1.5 or estimated creatinine clearance less than 40mL/min on baseline laboratory data.
* Clinically significant perianal fistulae
* Patients with diverting or end ostomy.
* Experimental therapy for Crohn's disease in the 4 weeks prior to study entry
* Presence of medical condition or disease that, in the opinion of the investigators, may place the patient at unacceptable risk for study participation, including, but not limited to, pregnancy, lactation, and/or inability/unwillingness to adhere to a contraceptive regimen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-10; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome will be clinical benefit which will be defined as a decrease in HBI, fecal lactoferrin, CRP and/or ESR at 6 weeks compared with baseline values | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Behm, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States